CLINICAL TRIAL: NCT06106984
Title: Home-based Rehabilitation Intervention for Phantom Limb Pain in Veterans With Lower Limb Amputations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B4805-W
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Phantom Limb Pain
Keywords: Amputation; Rehabilitation; Phantom limb pain; Pain
MeSH Terms: conditions — Phantom Limb; Pain

STUDY DESIGN:
Intervention Model Description: The investigators will conduct pilot testing of serial sessions of Graded Motor Imagery with Veterans using telehealth to their home environment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Veterans will trial the Graded Motor Imagery mobile application.
  Interventions: Device: Graded motor imagery mobile app

INTERVENTIONS:
Device: Graded motor imagery mobile app — The Graded Motor Imagery mobile app is a mobile app designed for intervention in phantom limb pain.

SUMMARY:
Nearly 60-85% of Veterans with amputations experience pain at the location of the amputated limb called phantom limb pain (PLP). PLP is a major problem and can have a profound impact on Veteran's daily function and ability to fully participate in life. Although several rehabilitation interventions are promising, advances in novel rehabilitation interventions are limited. The objective of this project is to refine a mobile app for graded motor imagery in 12 Veterans with amputations and test the mobile app with 36 Veterans with amputations. For this pilot project, the investigators will measure the preliminary feasibility and acceptability of the intervention. Knowledge from this project will provide evidence to guide future larger studies of this graded motor imagery intervention. Developing novel strategies for chronic pain in this population will positively impact quality of life for Veterans with amputations.

DETAILED DESCRIPTION:
Background: Phantom Limb Pain (PLP) is a form of unpredictable neuropathic pain in Veterans with amputation. Current non-medication treatments for PLP are limited and more interventions are needed that take into consideration the unique needs of the Veteran population. PLP significantly impairs rehabilitation outcomes and community participation. One non-medication intervention is graded motor imagery (GMI). GMI consists of sequentially progressing from limb laterality training, to motor imagery, and then mirror therapy (i.e., observing movement using the visual illusion of an intact limb in a mirror). Although clinicians report benefit from use of the technique, barriers exist to supporting at-home use of the intervention.

Research Questions (Objectives) - This VA Career Development Award-2 proposal focuses on refining a mobile app for GMI (VA-GMI) (Aim 1) and then pilot testing serial sessions of mobile app use in a sample of Veterans with lower limb amputation and moderate to severe PLP in their home setting (Aim 2).

Relevance to VA - There is a growing population of Veterans with amputation in the VA system. Many of whom will experience amputation pain, like phantom limb pain, and other amputation-related experiences. There are currently limited non-drug treatment options for phantom limb pain. Graded Motor Imagery could be one tool as a part of a comprehensive treatment plan for phantom limb pain. With the support of the expert mentor team in place, this work will incorporate Veteran input into the design of a novel intervention with high translational value. This work will lead to future investigations of optimized GMI intervention for the reduction of PLP in Veterans with amputations.

Number of Research Participants (Sample Size) - For Aim 1 that involves refining the mobile app, the investigators will recruit 12 Veterans. For Aim 2 that involves the clinical trial, the investigators will recruit 36 Veterans with unilateral below knee amputation to participate in the pilot testing of serial sessions.

Participating Sites - Minneapolis VA Health Care System

Duration of Participant Intake (Study Duration) - This project is projected to occur over 5 years. This project will begin with a 1 year refinement of the investigators' Graded Motor Imagery mobile app with 12 Veterans with amputation and moderate to severe PLP. In years 2-5, the investigators will conduct a pilot study to evaluate the feasibility and acceptability of the intervention with 36 Veterans with amputation and moderate to severe PLP. The investigators will conduct this study virtually with all Veterans in their home environment. All Veterans will receive twelve intervention sessions. Recruitment will conclude with 6-months remaining in the study timeline, which will be used for the dissemination of results and closure of the project.

Treatment (follow-up) - The Veterans in the pilot study will have 12 sessions of Graded Motor Imagery using the mobile app. The investigators will then follow Veterans for 3 and 6 month follow ups to learn more about their perspective of the Graded Motor Imagery mobile app.

Endpoints - The primary outcomes for this study are acceptability (Acceptability of Intervention Measure) and secondary measures of health outcomes, specifically pain interference (Amputation Related Pain and Experiences).

Qualitative Data - In addition to measuring acceptability and pain interference, the investigators will conduct semi-structured interviews with participants to develop further understanding of the benefits and drawbacks of Graded Motor Imagery in the home setting, using the mobile app.

ELIGIBILITY:
Inclusion Criteria:

* Must be a military Veteran
* At least 18 years old;
* >1 year since unilateral below knee amputation;
* Moderate or severe (NRS score 4 on a 0-10 scale) PLP;
* Stable medications over the past 2 weeks;
* Willing and able to give informed consent; and
* Able to participate in the telehealth study activities with a personal device.

Exclusion Criteria:

* Unstable medical conditions (e.g., uncontrolled diabetes, heart failure exacerbation);
* Unstable mental illness or substance use disorder (e.g., active suicidality or psychosis); and
* Unable to give informed consent due to a cognitive impairment.
* Fibromyalgia or complex regional pain syndrome-like symptoms

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure | 6-week post-test
  The Acceptability of Intervention Measure is a measure of the acceptability of the intervention sessions and if acceptability changes over time. This measure will evaluate the acceptability of using a mobile app with a telehealth platform. Minimum score: 12, maximum score: 60. A higher score indicates greater acceptability of the intervention, a lower score indicates lower acceptability of the intervention.
Change from 6-week post-test on the Acceptability of Intervention Measure to 6 months | 6 month follow up (an average of 24 weeks from 6-week post test)
  The Acceptability of Intervention Measure is a measure of the acceptability of the intervention sessions and if acceptability changes over time. This measure will evaluate the acceptability of using a mobile app with a telehealth platform. Minimum score: 12, maximum score: 60. A higher score indicates greater acceptability of the intervention, a lower score indicates lower acceptability of the intervention.

SECONDARY OUTCOMES:
Change from baseline Amputation Related Pain and Experiences to 6-weeks (post-test) | Baseline, 6-week Post-Test
  The Amputation Related Pain and Experiences is a measure to differentiate types of amputation-related pain and measure intensity, frequency, and pain interference with residual limb, phantom sensation, and phantom limb pain. For each section of residual limb pain, phantom sensation, and phantom limb pain, the minimum score is 0 and the maximum score is 60. A higher score indicates greater pain or sensation in each of the categories and a lower score indicates lower pain or sensation in each of the categories.
Change from 6-week post-test on the Acceptability of Intervention Measure at 3 months | 3 month follow up (an average of 12 weeks after baseline)
  The Acceptability of Intervention Measure is a measure of the acceptability of the intervention sessions and if acceptability changes over time. This measure will evaluate the acceptability of using a mobile app with a telehealth platform. Minimum score: 12, maximum score: 60. A higher score indicates greater acceptability of the intervention, a lower score indicates lower acceptability of the intervention.
Change from 6-week post-test Amputation Related Pain and Experiences to 3 months | Baseline, 3 month follow up (an average of 12 weeks from baseline)
  The Amputation Related Pain and Experiences is a measure to differentiate types of amputation-related pain and measure intensity, frequency, and pain interference with residual limb, phantom sensation, and phantom limb pain. For each section of residual limb pain, phantom sensation, and phantom limb pain, the minimum score is 0 and the maximum score is 60. A higher score indicates greater pain or sensation in each of the categories and a lower score indicates lower pain or sensation in each of the categories.
Change from baseline Amputation Related Pain and Experiences to 6 months | Baseline, 6 month follow up (an average of 24 weeks from baseline)
  The Amputation Related Pain and Experiences is a measure to differentiate types of amputation-related pain and measure intensity, frequency, and pain interference with residual limb, phantom sensation, and phantom limb pain. For each section of residual limb pain, phantom sensation, and phantom limb pain, the minimum score is 0 and the maximum score is 60. A higher score indicates greater pain or sensation in each of the categories and a lower score indicates lower pain or sensation in each of the categories.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya L Rich, PhD MA BS, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No